CLINICAL TRIAL: NCT00565110
Title: Effectiveness Study of a Stepped Care Depression Algorithm for Patients With Cancer
Brief Title: Treating Depression Among Low-Income Patients With Cancer
Acronym: ADAPt-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathleen R. Ell, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USCIRB-HS-10-00466; R01CA105269 (NIH)
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Major Depression; Dysthymia
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (No Intervention): EUC patients receive medical center standard oncology care and supportive services routinely provided to all patients with cancer. In addition, EUC patients are given a patient focused and a family focused educational pamphlet on depression and cancer and a listing of financial and community resources (in Spanish for Spanish-speaking patients). With patient consent, as described in the informed written consent, the treating oncologist is informed via medical chart note if EUC patients screen positive for major depression. Treating oncology attending physicians, fellows and residents are invited to attend a didactic session led by the study psychiatrist on treating depression in cancer patients.
- ADAPt-C intervention (Experimental): Intervention patients receive: first-line choice of antidepressant medication management,psychotherapy or both; depression education, and maintenance/relapse prevention counseling based on a stepped care depression treatment algorithm, treatment follow-up and feedback to the oncologist, and systems navigation; a psychiatric consultant who prescribes antidepressant medication for individual patients; and a didactic for oncologists on depression management. Cultural adaptations include: patient choice of first line treatment and degree of family participation in their depression care; PST tailored for literacy and patients with cancer; bilingual, bicultural CDCS; Spanish educational materials.
  Interventions: Behavioral: ADAPt-C intervention

INTERVENTIONS:
Behavioral: ADAPt-C intervention — Experimental Arm patients receive: first-line choice of antidepressant medication management,psychotherapy or both; depression education, and maintenance/relapse prevention counseling based on a stepped care depression treatment algorithm, treatment follow-up and feedback to the oncologist, and systems navigation; a psychiatric consultant who prescribes antidepressant medication for individual patients; and a didactic for oncologists on depression management. Cultural adaptations include: patient choice of first line treatment and degree of family participation in their depression care; PST tailored for literacy and patients with cancer; bilingual, bicultural CDCS; Spanish educational materials.
  Arms: ADAPt-C intervention

SUMMARY:
The ADAPt-C collaborative depression care model is designed to: improve depression symptom reduction in the intervention group over the modestly enhanced usual care group of low-income, predominantly Hispanic, patients with cancer who are receiving care in an urban public sector care system; and to improve quality of life outcomes among intervention patients over enhanced usual care.

DETAILED DESCRIPTION:
This controlled trial has tested the effectiveness of a socio-culturally tailored depression care program that includes a patient-centered approach to antidepressant medication management or structured psychotherapy (Problem Solving Treatment (PST)), patient/family depression education, treatment maintenance and relapse prevention counseling. Intervention enhancements include: depression care management based on a stepped care depression treatment algorithm; extension of the oncology care management team with a master's degreed social worker, who acts as Cancer Depression Clinical Specialist (CDCS) and provides PST, treatment follow-up and feedback to the oncologist, and who facilitates patient-provider communication and health system and community resources navigation; a psychiatric consultant, who provides supervision of the CDCS and consultation and antidepressant medication prescription for individual patients; and a didactic for oncologists on depression management. Cultural sensitivity and competency enhancements include: patient choice of first line treatment (antidepressant medication/PST) and degree of family participation in their depression care; PST tailored for language and literacy of patients with cancer; bilingual, bicultural CDCS; Spanish educational materials; and communication facilitation. Enhanced Usual Care (EUC) patients will receive the care and services routinely provided patients with cancer plus an educational/resource pamphlet for patients and for family members(on depression and cancer, depression treatment, talking with your doctor about your depression, and medical center and community mental health care resources). With patient consent, the oncologist is informed if EUC patients screen positive for major depression/dysthymia.

ELIGIBILITY:
Inclusion Criteria:

- 90 days post cancer diagnosis receiving acute cancer treatment or active follow-up

Exclusion Criteria:

- patients with advanced cancer or another medical condition that limited life expectancy to less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen R Ell, DSW, Principal Investigator — University of Southern California, School of Social Work
Locations (1):
- Los Angeles County+University of Southern California Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
National Cancer Institute, "Project ADAPT-C" selected for Research-Tested Interventions NCI Program 2014, http://rtips.cancer.gov/rtips/programDetails.do?programId=3551008. https://researchtoreality.cancer.gov/featured-r2r-partners/kathleen-ell-dsw
  1. ADAPt-C randomized clinical trial selected by the Predicting OptimaL cAncer RehabIlitation and Supportive care (POLARIS Consortia) led by the Netherlands

REFERENCES:
- [Background] Ell K, Quon B, Quinn DI, Dwight-Johnson M, Wells A, Lee PJ, Xie B. Improving treatment of depression among low-income patients with cancer: the design of the ADAPt-C study. Gen Hosp Psychiatry. 2007 May-Jun;29(3):223-31. doi: 10.1016/j.genhosppsych.2007.01.005. PMID 17484939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Usual Care | ADAPt-C Intervention
Started | 230 | 242
12-Month | 114 | 144
Completed | 99 | 111
Not Completed | 131 | 131

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | ADAPt-C Intervention | Total
Number analyzed (Participants) | 230 | 242 | 472
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.77 (12.93) | 47.59 (12.88) | 48.65 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 202 | 399
  Male | 33 | 40 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 196 | 219 | 415
  Not Hispanic or Latino | 34 | 23 | 57
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 230 | 242 | 472

OUTCOME MEASURES:

1. Primary Outcome: Reduced Depression Symptoms
Description: Number of participants with 50% PHQ-9 score reduction since baseline
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | ADAPt-C Intervention
Number analyzed (Participants) | 114 | 144
Participants | 57 | 91

2. Secondary Outcome: Physical Composite Summary Score (PCS) Derived From the 12-item Short Form (SF-12) Health Survey
Description: The SF-12 measures 8 health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. PCS is a summary score measuring physical health derived by summing responses across scale items and then transforming to a 0-100 scale (higher scores indicate better health).
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Enhanced Usual Care | ADAPt-C Intervention
Number analyzed (Participants) | 114 | 144
units on a scale | 38.68 (0.91) | 41.48 (0.84)

ADVERSE EVENTS:
Time Frame: 2 years
Description: The study intervention provided only behavioral sessions, thus no serious and other non-serious adverse events were collected or assessed systematically. However, we documented event information revealed by family member of participants, if any.
Arm/Group | Enhanced Usual Care | ADAPt-C Intervention
All-Cause Mortality (participants affected / at risk) | 54/230 | 45/242
Serious Adverse Events (participants affected / at risk) | 55/230 | 47/242
Other Adverse Events (participants affected / at risk) | 0/230 | 0/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care (N=230) | ADAPt-C Intervention (N=242)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 54 (54) | 45 (45) — event revealed by family member
In hospice or palliative care (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) — event revealed by family member

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No